CLINICAL TRIAL: NCT07335094
Title: A Clinical Study of Humanized CD19 CAR-T Cells With TLR2 for the Treatment of Adult Patients With Naive B-Cell Acute Lymphoblastic Leukemia/Lymphoma Who Are Intolerant to Intensive Chemotherapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Li Yuhua, professor, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024LX0089_GY
Record Dates: First submitted 2026-01-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: B Lymphoblastic Leukemia/Lymphoma
Keywords: CAR-T; CD19
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Administer a single infusion of humanized CD19 CAR-T Cells with TLR2 to this group of patients following fludarabine plus cyclophosphamide (F+C) lymphodepletion, and conduct follow-up surveys at the required time points within three years post-infusion according to the visit schedule.
  Interventions: Biological: humanized CD19 CAR-T Cells with TLR2

INTERVENTIONS:
Biological: humanized CD19 CAR-T Cells with TLR2 — Administer a single infusion of humanized CD19 CAR-T Cells with TLR2 to this group of patients following fludarabine plus cyclophosphamide (F+C) lymphodepletion

SUMMARY:
The purpose of this clinical trial is to tolerability and safety of humanized CD19 CAR-T therapy with TLR2 in adult patients with acute B lymphoblastic leukemia/lymphoma who cannot tolerate intense chemotherapy at initial treatment. Participants will receive a single infusion of CD19 CAR-T and complete follow-ups over the next three years.

DETAILED DESCRIPTION:
Objective: To evaluate the tolerability and safety of humanized CD19 CAR-T therapy with TLR2 in adult patients with acute B lymphoblastic leukemia/lymphoma who cannot tolerate intense chemotherapy at initial treatment. Secondary objective: To evaluate the efficacy and cytodynamics of humanized CD19 CAR-T therapy with TLR2 in adult acute B lymphoblastic leukemia/lymphoma who cannot tolerate intense chemotherapy at initial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly treated patients with acute B-lymphocytic leukaemia/lymphoma who are clinically determined to be unable to tolerate strong chemotherapy;
2. age 18-80 years old (including boundary value), both men and women can;
3. The physical status of the American Eastern Cancer Collaboration Group (ECOG) was 0~2 points;
4. Positive CD19 confirmed by flow cytometry and/or histopathology;
5. The expected survival period from the date of signing the informed consent form is more than 3 months.；
6. women of childbearing age screening period human chorionic gonadotropin (HCG) test negative, and Consent to use contraception for at least 1 year after the infusion; A man whose partner is fertile Subjects must agree to use an effective barrier contraceptive method for at least 1 year after the infusion；
7. the patient's main tissues and organs function well: (1) Liver function: ALT/AST<3 times the upper limit of normal (ULN) and total bilirubin ≤34.2μmol/L; (2) Renal function: creatinine clearance (Cockcroft-Gault method) ≥60mL/min; (3) Lung function: blood oxygen saturation ≥95%, and no active lung infection; (4) Cardiac function: left ventricular ejection fraction (LVEF) ≥50%; No large number of pericardium was found Fluid accumulation, no clinically significant electrocardiogram abnormalities；

Exclusion Criteria:

1. severe cardiac insufficiency, left ventricular ejection fraction <50%;
2. have a history of severe lung function impairment;
3. Combined with other advanced malignant tumors;
4. Had severe infection within 4 weeks before enrollment and could not be effectively controlled;
5. suffering from serious autoimmune diseases or immune deficiency diseases;
6. active hepatitis (HBV DNA quantitative > 500IU/ml] or HCV ribose Nucleic acid [HCVRNA] test positive);
7. human immunodeficiency virus (HIV) infection or known to have acquired immunodeficiency syndrome Co-syndrom (AIDS), or syphilis infection;
8. Have a history of severe allergy to biological products (including antibiotics), antibodies or cytokines Allergy to macromolecular biological drugs;
9. Acute graft-versus-host reactions were still present one month after immunosuppressant discontinuation Patients with allogeneic hematopoietic stem cell transplantation (GvHD);
10. in the pregnancy period (urine/blood pregnancy test positive) or breastfeeding women; nearly Men or women who plan to conceive within 1 year; Not guaranteed to be taken within 1 year after enrollment Effective contraception (condoms or contraceptives, etc.);
11. History of clinically significant central nervous system diseases, such as epilepsy, paresis, and loss Speech, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic Cerebral syndrome;
12. Suffering from mental illness;
13. The patient has substance abuse/addiction;
14. Use of banned drugs. (1). Hormones: within 7 days before leukocyte collection, or within 72 hours before CD19CAR-T administration A past therapeutic dose of corticosteroid (defined as prednisone or equivalent > 20mg/day) Days). However, the use of physiological substitutes, topical and inhaled steroids is permitted. (2) Chemotherapy: rescue chemotherapy was received within 2 weeks before white blood cell collection. (3) Allogeneic cell therapy: donor lymphocytes were received within 4 weeks before white blood cell collection Infusion. (4).GVHD treatment: Anti-GVHD received within 4 weeks prior to CD19CAR T cell infusion Heal. (5) Alenzumab was used within 6 months before white blood cell collection, or chlorine was used within 3 months Farabine or cladobine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  Objective response rates (ORR), including CR and PR, were analyzed by Clopper-Pearson distribution with bilateral 95% confidence intervals. For progression-free survival (PFS), Kaplan-Meier method was used to estimate the survival curve. Overall survival: the time from cell retransfusion until death from any cause.

IPD SHARING:
Plan to Share IPD: No